CLINICAL TRIAL: NCT03449589
Title: Effect of Smoking on Pain and Atherosclerosis in Patients With Rheumatoid Arthritis
Acronym: RAsmo
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: RÖK
Record Dates: First submitted 2018-02-07; First posted 2018-02-28 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Atherosclerosis; Pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Atherosclerosis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smokers: RA patients currently smoking
- Former smokers: RA patients who previously smoked
- Non smokers: Non smoking RA patients

SUMMARY:
Primary aim: examine a possible connection between cigarette smoking, disease activity and perceived pain in patients with rheumatoid arthritis.

Secondary aim: Evaluate cardiovascular risk in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
The study will recruit patients with rheumatoid arthritis (age 20-60 years) at rheumatology clinics in Västra Götaland. All patients meeting the inclusion criteria will be informed of the study in a letter and later contacted by the study coordinator and if interested booked for a study visit at the rheumatology clinic. At the study visit the patients will meet with rheumatologist for clinical examination of their joints and tenderpoints. An algometer is used for objective quantification of the patients pain sensitivity. Questionnaire regarding medical treatment, other diseases, smoking habits, subjective pain, fatigue, anxiety and depression, ability to work and ability to perform everyday activities are filled out by the patient.

Height, weight, blood pressure, blood, urine and fat biopsy will be collected for analyse.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-60 years diagnosed with rheumatoid arthritis

Exclusion Criteria:

* Other serious physical or mental illness, lack of knowledge in Swedish language making answering the questionnaires impossible

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Rheumatoid arthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Disease activity score (DAS 28) | At patient enrollment/study visit
  Difference in disease activity score (DAS 28) in smoking vs non-smoking RA-patients
  Disease activity, DAS28, is calculated using a specific formula based on:
  number of painful joints out of 28 joints examined number of swollen joints out of 28 joints examined erythrocyte sedimentation rate (ESR) or C reactive protein (CRP) patient's global assessment of disease activity on a 100 mm visual analogue scale (VAS)
  DAS thresholds:
  DAS28 lower than 2.6: remission DAS28 below 3.2: low disease activity DAS28 over 3.2 and under 5.1: moderate disease activity DAS28 above 5.1: high disease activity
Pain sensitivity (Pressure Pain Detection Threshold, PPDT) | At patient enrollment/study visit
  Difference in pain sensitivity in smoking vs non-smoking RA-patients. Testing of of all patients' pressure pain detection threshold (PPDT), i-e pain sensitivity is performed by trained personnel, using an algometer. The algometer is placed bilaterally on the nail of the thumb and on the second metatarsophalangeal joint (MTP2), giving a total of four measured points. A progressively increasing pressure is applied with the algometer and the patients are carefully instructed to signal as soon as the pressure sensation turns into pain (not to withstand the pain) and the algometer is removed. The amount of applied force shown in kPa in the display is reported as the PPDT. The measurements are performed twice for each point and an average value is calculated as the patients' pain sensitivity threshold/pressure pain detection threshold.
Subjective pain perception (VAS) | At patient enrollment/study visit
  Difference in pain perception in smoking vs non-smoking RA-patients
  Subjective pain perception is registered by self-reported estimation of pain on a visual analogue scale (VAS) of 100 mm concerning the week preceding the study.
Cardiovascular risk | At patient enrollment/study visit
  Difference in cardiovascular risk (Framingham score) in smoking vs non-smoking RA-patients
  The Framingham risk score is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual calculated on the basis of the following:
  Age Gender Total cholesterol HDL cholesterol Smoker Diabetes Systolic blood pressure Treatment for high blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Rheumatology and Inflammation research, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erlandsson MC, Malmhall-Bah E, Chandrasekaran V, Andersson KME, Nilsson LM, Toyra Silfversward S, Pullerits R, Bokarewa MI. Insulin Sensitivity Controls Activity of Pathogenic CD4+ T Cells in Rheumatoid Arthritis. Cells. 2024 Dec 22;13(24):2124. doi: 10.3390/cells13242124. PMID 39768214
- [Derived] Lyngfelt LI, Erlandsson MC, Nadali M, Hedjazifar S, Pullerits R, Andersson KM, Brembeck P, Silfversward ST, Smith U, Bokarewa MI. Impact of the Uncoupling Protein 1 on Cardiovascular Risk in Patients with Rheumatoid Arthritis. Cells. 2021 May 7;10(5):1131. doi: 10.3390/cells10051131. PMID 34067093
- [Derived] Nadali M, Lyngfelt L, Erlandsson MC, Silfversward ST, Andersson KME, Bokarewa MI, Pullerits R. Low Soluble Receptor for Advanced Glycation End Products Precedes and Predicts Cardiometabolic Events in Women With Rheumatoid Arthritis. Front Med (Lausanne). 2021 Jan 28;7:594622. doi: 10.3389/fmed.2020.594622. eCollection 2020. PMID 33585503